CLINICAL TRIAL: NCT00255710
Title: Nonmyeloablative Bone Marrow Transplants in Hematologic Malignancies: Dose Finding Study for Post-Transplant Immunosuppression
Brief Title: Cyclophosphamide and/or Mycophenolate Mofetil With or Without Tacrolimus in Treating Patients Who Are Undergoing a Donor Bone Marrow or Peripheral Stem Cell Transplant for Hematologic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000449652; P01CA015396 (NIH); P30CA006973 (NIH); JHOC-J0169; WIRB-20020304
Record Dates: First submitted 2005-11-18; First posted 2005-11-21 (Estimated); Last update posted 2010-03-17 (Estimated); Status verified 2010-03

CONDITIONS: Chronic Myeloproliferative Disorders; Graft Versus Host Disease; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Diseases
Keywords: graft versus host disease; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; chronic idiopathic myelofibrosis; chronic myelomonocytic leukemia; chronic phase chronic myelogenous leukemia; myelodysplastic/myeloproliferative disease, unclassifiable; previously treated myelodysplastic syndromes; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; stage II multiple myeloma; stage III adult Hodgkin lymphoma; stage III chronic lymphocytic leukemia; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III multiple myeloma; stage III small lymphocytic lymphoma; stage IV adult Hodgkin lymphoma; stage IV chronic lymphocytic leukemia; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV small lymphocytic lymphoma; stage II mycosis fungoides/Sezary syndrome; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; refractory anemia with excess blasts in transformation; refractory anemia with excess blasts; refractory cytopenia with multilineage dysplasia; primary systemic amyloidosis; de novo myelodysplastic syndromes; secondary acute myeloid leukemia; secondary myelodysplastic syndromes; atypical chronic myeloid leukemia
MeSH Terms: conditions — Myeloproliferative Disorders; Graft vs Host Disease; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Congenital Abnormalities; Primary Myelofibrosis; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic-Phase; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Hodgkin Disease; Leukemia, Lymphocytic, Chronic, B-Cell; Mycosis Fungoides; Sezary Syndrome; Anemia, Refractory, with Excess of Blasts; Immunoglobulin Light-chain Amyloidosis; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative | interventions — Filgrastim; Cyclophosphamide; fludarabine phosphate; Mycophenolic Acid; Tacrolimus; Peripheral Blood Stem Cell Transplantation; Radiotherapy

INTERVENTIONS:
Biological: filgrastim
Drug: cyclophosphamide
Drug: fludarabine phosphate
Drug: mycophenolate mofetil
Drug: tacrolimus
Procedure: allogeneic bone marrow transplantation
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Giving low doses of chemotherapy, such as fludarabine, and radiation therapy before a donor bone marrow or stem cell transplant helps stop the growth of cancer cells. It also stops the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune system and help destroy any remaining cancer cells (graft-versus-tumor effect). Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving cyclophosphamide, mycophenolate mofetil, and tacrolimus after transplant may stop this from happening.

PURPOSE: This phase I trial is studying cyclophosphamide and/or mycophenolate mofetil with or without tacrolimus to see which is the best regimen in treating patients who are undergoing a donor bone marrow or stem cell transplant for hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine a minimal (short-duration) post-transplant immunosuppression regimen comprising cyclophosphamide and/or mycophenolate mofetil with or without tacrolimus that results in ≤ 20% incidence of grade II or higher acute graft-versus-host disease (GVHD) in patients with hematologic malignancies undergoing nonmyeloablative allogeneic bone marrow or peripheral blood stem cell transplantation from an HLA-identical related donor.
* Determine the post-transplant immunosuppression regimen that results in < 10% incidence of nonengraftment, defined as < 5% donor chimerism in peripheral blood at day 60, in these patients.
* Determine the incidence and severity of acute GVHD in patients treated with these regimens.
* Determine the frequency of mixed chimerism in patients treated with these regimens.

OUTLINE:

* Nonmyeloablative allogeneic bone marrow transplantation (BMT) or peripheral blood stem cell transplantation (PBSCT): Patients receive fludarabine IV on days -4 to -2 and undergo total-body irradiation on day -1. Patients undergo allogeneic BMT on day 0 or PBSCT on day 0 (and days 1 and 2, if needed). Patients receive filgrastim (G-CSF) beginning on day 5 and continuing until at least day 15 or until blood counts recover.
* Sequentially increasing levels of post-transplant immunosuppression: Cohorts of patients are enrolled into 1 of the following regimens:

  * Regimen 1 (post-BMT immunosuppression): Patients receive cyclophosphamide IV on day 3 only.
  * Regimen 2 (post-BMT immunosuppression): Patients receive mycophenolate mofetil (MMF) once on day 3 and then twice daily on days 4-32.
  * Regimen 3 (post-BMT immunosuppression): Patients receive cyclophosphamide IV on days 3 and 4 and MMF twice daily on days 4-33.
  * Regimen 4 (post-PBSCT immunosuppression): Patients receive cyclophosphamide and MMF as in regimen 3.
  * Regimen 5 (post-PBSCT immunosuppression): Patients receive cyclophosphamide and MMF as in regimen 3 and tacrolimus twice daily on days 4-33.

Cohorts of approximately 10-20 patients receive sequentially increasing levels of post-transplant immunosuppression until a minimal (short-duration) post-transplant immunosuppression regimen is identified. The minimal post-transplant immunosuppression regimen is defined as the regimen in which ≤ 3 of 10 or ≤ 6 of 20 patients develop grade II or higher acute graft-versus-host disease AND ≤ 2 of 10 or ≤ 4 of 20 patients fail to engraft 60 days post-transplantation. Once the minimal post-transplant immunosuppression regimen is identified, an additional 10 patients are treated with that regimen.

Patients are followed for 60 days after transplantation.

PROJECTED ACCRUAL: A total of 60 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following hematologic malignancies:

  * Stage II or III multiple myeloma
  * Amyloidosis
  * Myelofibrosis with ≥ 2 of the following high-risk features:

    * Over 55 years of age
    * Hemoglobin < 10 g/dL
    * WBC < 3,000/mm^3 OR > 10,000/mm^3
    * Platelet count < 100,000/mm^3
    * Cytogenetic abnormalities
  * Mycosis fungoides, meeting 1 of the following criteria:

    * Stage IIB or III disease with evidence of histologic conversion to an aggressive lymphoma

      * Must demonstrate chemosensitivity
    * Stage IV disease
  * Paroxysmal nocturnal hemoglobinuria

    * Not meeting criteria for other bone marrow transplantation (BMT) or treatment studies
  * Diagnosis of 1 of the following hematologic malignancies, for which patient is not eligible for potentially curative allogeneic BMT due to end-organ dysfunction, age 65 to 75, or the amount of prior chemotherapy:

    * Acute myeloid or acute lymphoblastic leukemia

      * High-risk disease in first or second (or further) complete remission
    * Relapsed aggressive non-Hodgkin's lymphoma

      * Not eligible for autologous or standard allogeneic BMT
    * Hodgkin's lymphoma in second or further complete or partial remission

      * Not eligible for autologous or standard allogeneic BMT
    * Myelodysplastic syndromes or myelodysplastic/myeloproliferative diseases

      * Any of the following subtypes:

        * Refractory anemia with excess blasts (RAEB)
        * RAEB in transformation
        * Chronic myelomonocytic leukemia
        * Any morphologic subtype with multiple chromosomal abnormalities
        * Any subset with life-threatening cytopenias in all 3 cell lines, defined as platelet count ≤ 20,000/mm^3, absolute neutrophil count ≤ 500/mm^3, and reticulocyte count ≤ 50,000/mm^3
      * Meets both of the following criteria:

        * Less than 20% blasts by bone marrow biopsy
        * Not eligible for standard allogeneic BMT
      * No refractory anemia with ringed sideroblasts
      * No 5q syndrome
    * Stage III or IV chronic lymphocytic leukemia

      * Not meeting criteria for other BMT studies
    * Chronic myelogenous leukemia in first or second chronic phase

      * Not meeting criteria for other BMT studies or treatment
    * Stage III or IV indolent small lymphocytic or follicular lymphoma

      * Not eligible for autologous or standard allogeneic BMT or other active protocols at Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
* Must have an HLA-identical related donor available

PATIENT CHARACTERISTICS:

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* See Disease Characteristics

Hepatic

* Bilirubin ≤ 3.0 mg/dL
* AST ≤ 175 U/L
* ALT ≤ 200 U/L

Renal

* Creatinine ≤ 3.0 mg/dL

Cardiovascular

* LVEF ≥ 30%

Pulmonary

* FEV_1 ≥ 40% predicted
* Forced vital capacity ≥ 40% predicted

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative

PRIOR CONCURRENT THERAPY:

Chemotherapy

* See Disease Characteristics

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2002-07

PRIMARY OUTCOMES:
Post-transplant immunosuppression regimen with ≤ 20% incidence of a grade II-IV graft-versus-host-disease (GVHD) and < 10% incidence of nonengraftment (< 5% donor chimerism) at day 60 following transplant
Incidence and severity of acute GVHD at day 60 following transplant
Frequency of mixed chimerism defined as any detectable donor cells at day 60 following transplant

CONTACTS AND LOCATIONS:
Overall Officials: Carol A. Huff, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States